CLINICAL TRIAL: NCT07256288
Title: A Single-Center, Double-Blind, Placebo-Controlled, Dose-Escalating Phase Ia Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Characteristics of EA5 in a Single Dose in Adult Healthy Subjects
Brief Title: A Phase Ia Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of EA5 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Lanyi Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: C-EA5-2301
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- EA5 90mg (Experimental): EA5 was administered intravenously.
  Interventions: Drug: EA5
- EA5 180mg (Experimental): EA5 was administered intravenously.
  Interventions: Drug: EA5
- EA5 360mg (Experimental): EA5 was administered intravenously.
  Interventions: Drug: EA5; Drug: Placebo
- EA5 720mg (Experimental): EA5 was administered intravenously.
  Interventions: Drug: EA5; Drug: Placebo
- EA5 1440mg (Experimental): EA5 was administered intravenously.
  Interventions: Drug: EA5; Drug: Placebo
- Placebo (Placebo Comparator): Placebo was administered intravenously.
  Interventions: Drug: EA5

INTERVENTIONS:
Drug: EA5 — All doses of EA5 were administered by IV infusion, using programmable IV infusion pump and IV sets with in-line filters.
Drug: Placebo — All doses of placebo were administered by IV infusion, using programmable IV infusion pump and IV sets with in-line filters.
  Arms: EA5 1440mg; EA5 360mg; EA5 720mg

SUMMARY:
This is a single-center, double-blind, placebo-controlled, dose-escalating Phase Ia clinical study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of a single dose of EA5 in healthy adult subjects.

DETAILED DESCRIPTION:
The study plans to enroll up to 28 subjects. Its primary purpose is to conduct a preliminary assessment of the exposure, safety, and pharmacokinetic profile of EA5 in humans, thereby informing the confirmation or adjustment of the formal trial design. The trial is structured into a pilot phase and a formal phase, encompassing a total of five planned dose cohorts: the pilot trial involves two dose groups (90 mg and 180 mg), each with 2 subjects receiving the active drug; the formal trial consists of three dose groups (360 mg, 720 mg, and 1440 mg), where participants are randomized in a 3:1 ratio (6 subjects receiving the active drug EA5 and 2 subjects receiving placebo per cohort), administered via intravenous (IV) infusion.A 57-day observation period was performed for safety, pharmacokinetic, and pharmacodynamic assessments after study drug administration. Antidrug antibody (ADA) levels were monitored in study participants for the duration of the 57-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 55 years (inclusive), regardless of gender.
* Body weight ≥50 kg (male) or ≥45 kg (female), and a body mass index (BMI) between 18 and 28 kg/m² (inclusive).
* Must have received the meningococcal polysaccharide vaccine MenACWY (containing serogroups A, C, W, and Y) at least two weeks prior to dosing.
* Subjects must be able to communicate effectively with the investigator and are expected to comply with the study procedures as defined in the protocol.
* Subjects must be in good general health, as judged by the investigator based on medical history, physical examination, vital signs, electrocardiogram (ECG), chest X-ray, abdominal ultrasound, and laboratory test results.
* Male subjects agree to use effective contraception (vasectomy, abstinence, or condom) from screening until 6 months after the final study intervention. Female subjects must have a negative blood pregnancy test at screening and baseline. Throughout the study and for 6 months thereafter, all subjects and their partners (if of childbearing potential) must use highly effective non-pharmacological contraception.
* Subjects must provide written informed consent voluntarily before any study-specific procedures are performed.
* Systolic and diastolic blood pressure must be within the normal range, or exhibit abnormalities deemed clinically insignificant by the investigator.

Exclusion Criteria:

* History of severe drug allergy; or a clear history of allergy and/or known allergy to the investigational product or any of its excipients, which in the opinion of the investigator, renders the subject unsuitable for participation in the study.
* Prior history of splenectomy.
* History of pulmonary tuberculosis.
* Congenital or acquired complement deficiency (e.g., hypocomplementemia).
* Any contraindication to antibiotic prophylaxis (e.g., beta-lactam antibiotics, ciprofloxacin) for meningococcal infection
* Positive test for hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, treponemal antibody (TP-Ab), or hepatitis B virus (HBV) surface antigen (HBsAg) at screening
* Presence of symptoms or a significant history of any major disease, including but not limited to cardiac, hepatic, renal, other acute or chronic gastrointestinal or respiratory diseases; hematological, endocrine, neurological, psychiatric disorders; or any other disease or physiological condition that could interfere with the interpretation of the study results.
* Participation in any clinical trial involving an investigational drug or medical device within 3 months prior to screening, or within 5 half-lives of the previous investigational drug prior to screening (whichever is longer)
* Blood loss or donation > 400 mL within 3 months prior to screening, or > 200 mL within 4 weeks prior to screening, or intention to donate blood during the study period
* Average cigarette smoking of ≥5 cigarettes per day within 3 months prior to the study
* Alcohol abuse or regular alcohol consumption exceeding 14 units per week within 6 months prior to screening (1 unit ≈ 360 mL beer, 45 mL 40% spirits, or 150 mL wine), or a positive alcohol breath test at screening.
* History of drug abuse or a positive urine drug screen at screening
* Undergone surgery or received blood or blood product transfusion within 1 month prior to screening。
* Administration of any live or live-attenuated vaccine within 1 month prior to the first dose。
* Use of any prescription drugs, over-the-counter medications, herbal medicines, or vitamins within 14 days or 5 half-lives (whichever is longer) prior to screening。
* Presence of any active infection (viral, bacterial, or fungal), including herpes zoster or herpes simplex, within 14 days prior to dosing.
* History of fever (≥38°C) within 7 days prior to the first dose.
* Female subjects who are pregnant or lactating, or who have engaged in unprotected sexual intercourse within 14 days prior to the study.
* Inability to complete the study for any other reason, or considered by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Baseline up to Day 57
  TEAEs were defined as AEs that occurred on or after the date and time of study drug administration, or those that first occurred before dosing but worsened in frequency or severity after study drug administration. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of EA5 | 30 minutes predose, 5 minutes, 1, 2, 6, 24, hours postdose, then at Days 3, 4, 8, 15, 29, 43, 57
  Blood samples were collected for analysis of Cmax
Time To Maximum Observed Serum Concentration (Tmax) of EA5 | 30 minutes predose, 5 minutes, 1, 2, 6, 24, hours postdose, then at Days 3, 4, 8, 15, 29, 43, 57
  Blood samples were collected for analysis of Tmax
Area Under The Serum Concentration Versus Time Curve From Time Zero To The Time of The Last Quantifiable Concentration (AUC0-t) of EA5 | 30 minutes predose, 5 minutes, 1, 2, 6, 24, hours postdose, then at Days 3, 4, 8, 15, 29, 43, 57
  Blood samples were collected for analysis of AUC0-t
Area Under The Serum Concentration Versus Time Curve From Time Zero (Dosing) To Infinity (AUCinf) of EA5 | 30 minutes predose, 5 minutes, 1, 2, 6, 24, hours postdose, then at Days 3, 4, 8, 15, 29, 43, 57
  Blood samples were collected for analysis of AUCinf
Terminal Elimination Rate Constant (λz) of Serum EA5 | 30 minutes predose, 5 minutes, 1, 2, 6, 24, hours postdose, then at Days 3, 4, 8, 15, 29, 43, 57
  Blood samples were collected for analysis of λz
Terminal Elimination Half-life (t½) of Serum EA5 | 30 minutes predose, 5 minutes, 1, 2, 6, 24, hours postdose, then at Days 3, 4, 8, 15, 29, 43, 57
  Blood samples were collected for analysis of t½
Total Clearance (CL) of EA5 | 30 minutes predose, 5 minutes, 1, 2, 6, 24, hours postdose, then at Days 3, 4, 8, 15, 29, 43, 57
  Blood samples were collected for analysis of CL
Percent Change From Baseline in Free Complement Component 5 (C5) | Baseline, Day 57
  Blood samples were collected for analysis of free C5 concentrations.
Percent Change From Baseline in Total Complement C5 | Baseline, Day 57
  Blood samples were collected for analysis of total C5 concentrations.
Percent Change From Baseline in determination of terminal complement activity in serum | Baseline, Day 57
  Blood samples were collected for analysis of determination of terminal complement activity
Percentage of Participants With Positive Anti-Drug Antibody (ADA) | Baseline up to Day 57
  lood samples were collected to evaluate antibody response through development of ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Professor, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No